CLINICAL TRIAL: NCT03113240
Title: Effects of Enteral Glutamine on Intestinal Permeability in Hospitalized Patients With Enteral Feeding in Intensive Care Unit
Brief Title: Trial of Enteral Glutamine on Intestinal Permeability in Critically Ill Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate Professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 311/4114
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness; Enteral Nutrition; Intestinal Permeability
Keywords: Glutamin; Enteral Nutrition; Intensive Care Unit; Intestinal Permeability
MeSH Terms: conditions — Critical Illness | interventions — glutamin-(asparagin-)ase; Glutamine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glutamin (Experimental): Intervention patients will be received enteral formula and glutamine 0.3 g/kg/day given via nasogastric tube as boluses q 4hrs.
  Interventions: Drug: Glutamin
- maltodextrin (Placebo Comparator): Control patients will be received enteral formula and maltodextrin mixed in with water and given via nasogastric tube as boluses q 4hrs.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Drug: Glutamin — Enteral Glutamine 0.3g/kg/day powdered glutamine to be mixed in with water and given via nasogastric tube q4 hrs.
  Other Names: L-glutamine
  Arms: Glutamin
Other: Maltodextrin — Maltodextrin mixed with water given via NG tube q 4 hours.
  Arms: maltodextrin

SUMMARY:
Glutamine-induced recovery in intestinal barrier function by reducing bacterial translocation was demonstrated in previous studies. In this trial, intensive care unit patients with enteral feeding will receive either enteral glutamine or maltodextrin as placebo for 10 days and the effects of the intervention on intestinal permeability will be assessed.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in general intensive care unit (ICU) in Tehran, Iran. After a full review of the inclusion and exclusion criteria and explanation of the risks and benefits of the study, written consent form will be completed. The participants are 60 eligible hospitalized patients with enteral feeding in ICU, aged ≥ 18 years. Intervention patients will be received 0.3 g/kg/day of glutamine along with enteral formula for 10days and control patients will be received maltodextrin along with enteral formula for 10 days. Patients will be evaluated for plasma endotoxin and plasma zonulin.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) admitted to ICU
* Start of study intervention within 48 hours after ICU admission
* Expected to require enteral nutrition for at least 72 hours aiming for full enteral nutrition and receive at least 80 percent of enteral formula during the first 48 hour
* Written informed consent of patient or written informed consent of legal representative

Exclusion Criteria:

* Enrollment in a related ICU interventional study
* Requiring other specific enteral nutrition for medical reason
* Death or Discharge before 5th day
* Having any contra-indication to receive enteral nutrition
* Pregnant patients or lactating with the intent to breastfeed
* BMI <18 or > 40.0 kg/m2
* Have life expectancy of <6 mo
* Patients who are moribond
* Liver cirrhosis- Child's class C liver disease
* Have seizure disorder requiring anticonvulsant
* History of allergy or intolerance to the study product components
* Receiving glutamine during two weeks before start study product
* Have other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma endotoxin concentration | baseline, Day 5, Day 10
  The levels of plasma endotoxin
Maximum plasma zonulin concentration | baseline, Day 5, Day 10
  The levels of plasma zonulin
Maximum plasma antiendotoxin IgG and Ig M concentration | baseline, Day 5, Day 10
  The levels of plasma antiendotoxin IgG and Ig M concentration

SECONDARY OUTCOMES:
Gastrointestinal complication | Day10
  abdominal distention, vomiting, diarrhea and constipation
Mortality in ICU | Day 10
  Mortality rate in ICU
Length of stay in ICU | Day 10
  Duration of stay in ICU
Severe sepsis | Day 10
  according to the American College of Chest Physicians and the Society of Critical Care Medicine

OTHER OUTCOMES:
Serum Glutamin | baseline, Day 5, Day 10
  The levels of serum Glutamin

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, MD, PhD, Study Chair — Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Shohada Tajrish Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rao R, Samak G. Role of Glutamine in Protection of Intestinal Epithelial Tight Junctions. J Epithel Biol Pharmacol. 2012 Jan;5(Suppl 1-M7):47-54. doi: 10.2174/1875044301205010047. No abstract available. PMID 25810794
- [Background] dos Santos Rd, Viana ML, Generoso SV, Arantes RE, Davisson Correia MI, Cardoso VN. Glutamine supplementation decreases intestinal permeability and preserves gut mucosa integrity in an experimental mouse model. JPEN J Parenter Enteral Nutr. 2010 Jul-Aug;34(4):408-13. doi: 10.1177/0148607110362530. PMID 20631386
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Kreymann KG, Berger MM, Deutz NE, Hiesmayr M, Jolliet P, Kazandjiev G, Nitenberg G, van den Berghe G, Wernerman J; DGEM (German Society for Nutritional Medicine); Ebner C, Hartl W, Heymann C, Spies C; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Intensive care. Clin Nutr. 2006 Apr;25(2):210-23. doi: 10.1016/j.clnu.2006.01.021. Epub 2006 May 11. PMID 16697087
- [Background] D'Souza R, Powell-Tuck J. Glutamine supplements in the critically ill. J R Soc Med. 2004 Sep;97(9):425-7. doi: 10.1177/014107680409700904. No abstract available. PMID 15340021